CLINICAL TRIAL: NCT05822947
Title: Blinding Assessment of Manual Therapy Interventions of the Back in Swiss Graduate Students: a Blinding Feasibility Randomized Controlled Trial
Brief Title: Blinding Assessment of Manual Therapy Interventions of the Back in Swiss Graduate Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cesar A Hincapié, DC PhD (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Cesar A Hincapié, DC PhD, Senior Scientist and Head of Musculoskeletal Epidemiology Research, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SENSATE Blinding
Record Dates: First submitted 2023-03-02; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Back Pain; Back Disorder; Back Pain, Low
Keywords: Methods; Manual therapy; Randomised trial; Back pain; Feasibility; Blinding assessment
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single centre, two-parallel group, blinding feasibility randomized controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding was the primary outcome of interest. That said, except for intervention providers, every role was, by protocol, blinded to intervention assignment.
  To maintain blinding of participants, candidate participants were formally invited to participate by email, with a study information form that masked the blinding feasibility objective.
  The intervention providers were kept in a separate room and could not be blinded but were asked not to disclose the intervention group or the nature of the control MT component to participants, outcome assessors, data analysts, and other members of the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active manual therapy (Experimental): Active manual therapy intervention involved mobilization of the lumbar paraspinal musculature. With participants laying prone on a chiropractic table, the intervention provider administered hand-reinforced circumferential movements to six focal areas, using continuous ischemic compression strokes, and adjusting the pressure to participants' tolerability.
  Interventions: Other: Active manual therapy
- Control manual therapy (Sham Comparator): Control MT intervention included light touch to six distal, broad areas of the thoracic region, with a synchronized breathing exercise.
  Interventions: Other: Control manual therapy

INTERVENTIONS:
Other: Active manual therapy — Soft tissue mobilization of the lumbar paraspinal musculature (3 to 4 minutes).
  Arms: Active manual therapy
Other: Control manual therapy — Light touch and a breathing exercise (3 to 4 minutes).
  Arms: Control manual therapy

SUMMARY:
There is marked uncertainty regarding the feasibility of achieving adequate blinding in randomized controlled trials of manual therapy. In other words, whether participants and outcome assessors can accurately perceive randomly assigned interventions is unclear. This feasibility trial was conducted as part of a doctoral epidemiology course at the University of Zurich, Switzerland. Within the practice-based context of the class and using a study population of healthy graduate students enrolled in the course, the investigators aimed to evaluate blinding of participants randomly assigned (similar to tossing a coin) to one of two manual therapy interventions (active versus control). The investigators also aimed to assess blinding among outcome assessors.

DETAILED DESCRIPTION:
Manual therapy remains a guideline-compliant, first-line therapeutic option for back pain. Yet, maintaining methodological quality in randomized controlled trials of manual therapy interventions poses challenges, particularly concerning: (a) The design of adequate 'sham' controls and (b) the blinding status of participants and outcome assessors. Optimal implementation of large-scale manual therapy trials requires testing the feasibility of control manual therapy interventions and effective blinding of participants and outcome assessors. Even when conducted in healthy populations and non-clinical settings, blinding feasibility trials remain an opportunity for methodological advancement in the field of manual medicine, and a research priority for unbiased treatment effect estimation in future trials.

The primary objective of this methodological trial was to quantitatively assess blinding feasibility among participants (graduate students enrolled in an epidemiology Ph.D. course) assigned to an active or control intervention immediately after a one-time intervention session. The secondary objective was to assess blinding feasibility among outcome assessors and explore factors influencing perceptions about intervention assignment among participants and outcome assessors. These two objectives contributed to obtaining valuable preliminary measures of blinding (blinding indices) for a future methodological blinding feasibility trial to be carried out in a real-world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* enrolled in a doctoral-level epidemiology course at the University of Zurich, Switzerland.

Exclusion Criteria:

* serious pathology (i.e., cancer, severe scoliosis, inflammatory disease, infection, cauda equina syndrome or progressive motor deficit)
* history of spine surgery
* obvious contraindication to manual therapy (i.e., spinal fracture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Blinding feasibility of participants, measured by the Bang blinding index. | Immediately after the one-time intervention session (study day 1).
  The Bang blinding index ranges from -1 to 1, with 0 representing satisfactory blinding. It can be interpreted as the proportion of participants correctly answering their allocated intervention within an intervention arm beyond chance. For the Bang BI, a score with an absolute value of ≤0.3 (i.e., -0.3 to 0.3) was deemed compatible with satisfactory blinding, although blinding scenarios (comparing blinding indices in active vs. control arms) were discussed.
  Participants were asked: "To which extent do you know which intervention you received?" and were given five possible answers: "I strongly believe I received the active intervention", "I somewhat believe I received the active intervention", "I somewhat believe I received the control intervention", "I strongly believe I received the control intervention", and "I do not know [whether I received the active or control intervention]".

SECONDARY OUTCOMES:
Blinding feasibility of participants, measured by the James blinding index. | Immediately after the one-time intervention session (study day 1).
  The James blinding index ranges from 0 (all correct responses) to 1 (all 'don't know' responses), where 0.5 corresponds to 50% of responses being correct, and 50% incorrect. Lack of satisfactory blinding may be claimed if the two-sided confidence interval of the James blinding index does not cover 0.5.
  Immediately after the intervention, participants rated their perception about received intervention on a five-point scale: "I strongly believe I received the active intervention", "I somewhat believe I received the active intervention", "I somewhat believe I received the control intervention", "I strongly believe I received the control intervention", and "I do not know [whether I received the active or control intervention]".
Blinding feasibility of outcome assessors, measured by the Bang blinding index. | Immediately after the one-time intervention session (study day 1).
  The Bang blinding index ranges from -1 to 1, with 0 representing satisfactory blinding. It can be interpreted as the proportion of outcome assessors who correctly answered the allocated intervention of participants within an intervention arm beyond chance.
  Outcome assessors were asked, "To which extent do you know which intervention (active intervention or control intervention) the patient received?" on a five-point scale: "I strongly believe that they received the active intervention," "I somewhat believe that they received the active intervention," "I somewhat believe that they received the control intervention," "I strongly believe that they received the control intervention," "I don't know [whether this participant received active or control intervention]."
Factors contributing to perceived intervention arm allocation among study participants. | Immediately after the one-time intervention session (study day 1).
  Factors contributing to perceived intervention arm allocation among study participants were explored with an open-ended free text question: "Please briefly explain your answer regarding the question above [question above: "To which extent do you know which intervention you received?"].
Factors contributing to perceived intervention arm allocation among outcome assessors. | Immediately after the one-time intervention session (study day 1).
  Factors contributing to perceived intervention arm allocation among outcome assessors were explored with an open-ended free text question: "Please briefly explain your answer regarding the question above [question above: "To which extent do you know which intervention (active intervention or control intervention) the patient received?"].
Blinding feasibility of outcome assessors, measured by the James blinding index. | Immediately after the one-time intervention session (study day 1).
  The James blinding index ranges from 0 (all correct responses) to 1 (all 'don't know' responses), where 0.5 corresponds to 50% of responses being correct, and 50% incorrect. Lack of satisfactory blinding may be claimed if the two-sided confidence interval of the James blinding index does not cover 0.5.
  Outcome assessors were asked, "To which extent do you know which intervention (active intervention or control intervention) the patient received?" on a five-point scale: "I strongly believe that they received the active intervention," "I somewhat believe that they received the active intervention," "I somewhat believe that they received the control intervention," "I strongly believe that they received the control intervention," "I don't know [whether this participant received active or control intervention]."

OTHER OUTCOMES:
Back function - self-reported flexibility, immediately before the one-time intervention session. | Immediately before the one-time intervention session (study day 1).
  Participants answered the question, "How would you rate your back flexibility at the moment?" (adapted from The International Fitness Scale [IFIS]). Possible answers (5-point scale) include "Very poor," "Poor," "Average," "Good," and "Very good."
Back function - self-reported flexibility, immediately after the one-time intervention session. | Immediately after the one-time intervention session (study day 1).
  Participants answered the question, "How would you rate your back flexibility at the moment?" (adapted from The International Fitness Scale [IFIS]). Possible answers (5-point scale) include "Very poor," "Poor," "Average," "Good," and "Very good."
Back function - self-reported ache, pain, discomfort in the upper back, immediately before the one-time intervention session. | Immediately before the one-time intervention session (study day 1).
  Ache, pain, discomfort in the upper back by asking, "During the past week, have you experienced ache, pain, discomfort in your upper back?". If answered "Yes," participants were asked to rate the degree of discomfort: "How uncomfortable do you feel with the ache, pain, or discomfort in your upper back?". These two questions were adapted from the Cornell Musculoskeletal Discomfort Questionnaire.
Back function - self-reported ache, pain, discomfort in the upper back, immediately after the one-time intervention session. | Immediately after the one-time intervention session (study day 1).
  Ache, pain, discomfort in the upper back by asking, "During the past week, have you experienced ache, pain, discomfort in your upper back?". If answered "Yes," participants were asked to rate the degree of discomfort: "How uncomfortable do you feel with the ache, pain, or discomfort in your upper back?". These two questions were adapted from the Cornell Musculoskeletal Discomfort Questionnaire.
Back function - self-reported ache, pain, discomfort in the lower back, immediately before the one-time intervention session. | Immediately before the one-time intervention session (study day 1).
  Ache, pain, discomfort in the lower back by asking, "During the past week, have you experienced ache, pain, discomfort in your lower back?". If answered "Yes," participants were asked to rate the degree of discomfort: "How uncomfortable do you feel with the ache, pain, or discomfort in your lower back?". These two questions were adapted from the Cornell Musculoskeletal Discomfort Questionnaire.
Back function - self-reported ache, pain, discomfort in the lower back, immediately after the one-time intervention session. | Immediately after the one-time intervention session (study day 1).
  Ache, pain, discomfort in the lower back by asking, "During the past week, have you experienced ache, pain, discomfort in your lower back?". If answered "Yes," participants were asked to rate the degree of discomfort: "How uncomfortable do you feel with the ache, pain, or discomfort in your lower back?". These two questions were adapted from the Cornell Musculoskeletal Discomfort Questionnaire.
Lumbar spine range of motion, immediately before the one-time intervention session. | Immediately before the one-time intervention session (study day 1).
  Maximum active total flexion and extension (0 to 100+ degrees) in standing position, measured with a validated mobile phone measuring device placed at the level of T12. Higher scores represent higher flexibility.
Lumbar spine range of motion, immediately after the one-time intervention session. | Immediately after the one-time intervention session (study day 1).
  Maximum active total flexion and extension (0 to 100+ degrees) in standing position, measured with a validated mobile phone measuring device placed at the level of T12. Higher scores represent higher flexibility.
Change in lumbar spine range of motion, difference between after and before intervention measurements. | Immediately before and after the one-time intervention session (study day 1).
  Change in maximum active total flexion and extension (0 to 100+ degrees) in standing position, measured with a validated mobile phone measuring device placed at the level of T12. Higher scores represent higher flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar A Hincapié, DC PhD, Principal Investigator — Balgrist University Hospital and University of Zurich
Locations (1):
- University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator will make supporting information available upon reasonable request without compromising the privacy of the graduate students enrolled in the doctoral-level course.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Supporting information will be available once the manuscript is published in a peer-reviewed journal. Supporting information will be available indefinitely.
Access Criteria: The principal investigator may request a brief description of the intended aims before sharing supporting information.

REFERENCES:
- [Derived] Munoz Laguna J, Nyantakyi E, Bhattacharyya U, Blum K, Delucchi M, Klingebiel FK, Labarile M, Roggo A, Weber M, Radtke T, Puhan MA, Hincapie CA. Is blinding in studies of manual soft tissue mobilisation of the back possible? A feasibility randomised controlled trial with Swiss graduate students. Chiropr Man Therap. 2024 Jan 29;32(1):3. doi: 10.1186/s12998-023-00524-x. PMID 38287417